CLINICAL TRIAL: NCT06163677
Title: Patient-Reported Outcomes Associated With COVID-19 and Influenza: A Prospective Survey Study on Outpatient Symptomatic Adults With Laboratory-Confirmed Illness in the United States
Brief Title: A Study to Look at the Health Outcomes of Patients With COVID-19 and Influenza.
Status: Withdrawn | Type: Observational
Why Stopped: Study cancelled due to change in feasibility.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591064
Record Dates: First submitted 2023-12-07; First posted 2023-12-11 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Coronavirus Disease 2019; Influenza
Keywords: Patient-Reported Outcomes; Humanistic Burden; Quality of Life; Disease Symptoms Assessment; COVID-19; SARS-CoV-2; Severe Acute Respiratory Syndrome Coronavirus 2 Infection; Acute respiratory infection; Influenza; Human Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive: Laboratory-confirmed COVID-19 illness and at least one patient-reported symptom
  Interventions: Biological: COVID-19 Vaccine
- Influenza Positive: Laboratory-confirmed influenza illness and at least one patient-reported symptom

INTERVENTIONS:
Biological: COVID-19 Vaccine — Receipt of Pfizer BioNTech COVID-19 vaccine
  Groups: COVID-19 Positive

SUMMARY:
The main purpose of this study is to understand:

* the symptoms of COVID-19 or influenza
* health-related outcomes of people with COVID-19 or influenza
* the effects of vaccines in people with COVID-19 or influenza.

This study will take in participants who are:

* 18 years or older
* reported to have symptoms with lab tests that have confirmed illness. The lab tests can be tested at any of Walgreens pharmacy COVID-19 or influenza test sites.

The study will collect vaccine history information from participants who are ready to take part in the study. Participant will be emailed a form with questions about their health related to COVID-19 or influenza during twelve follow-ups over a 6-month period.

DETAILED DESCRIPTION:
This is a prospective non-interventional longitudinal cohort survey study. Repeated measures on PROs: symptoms (prevalence, frequency, duration, and severity), EQ-5D-5L, WPAI and PROMIS-Fatigue short form 8a over 6 months will be collected and evaluated.

COVID-19 Cohort: Participants 18 years or older with laboratory-confirmed COVID-19 illness and at least one patient-reported symptom.

Influenza Cohort: Participants 18 years or older with laboratory-confirmed influenza illness and at least one patient-reported symptom.

All study objectives and outcomes will be assessed separately for the two study cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-reported at least one symptom in the screening questionnaire
* Positive result reported from the laboratory
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study
* Able to complete the questionnaires by themselves in English

Exclusion Criteria:

* Positive result for both COVID-19 and influenza (coinfection)
* COVID-19 test is done with non-RT-PCR methods such as a rapid antigen test or antibody test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants 18 years or older who are self-reported symptomatic, with laboratory-confirmed illness when tested at any of Walgreens pharmacy COVID-19 or influenza test sites, and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Prevalence, Severity, and duration of SARS-CoV-2 symptoms | 6 Months
  To characterize prevalence and duration of SARS-CoV-2 symptoms before COVID-19 and up to 6 months (acute phase and Long COVID).
Prevalence, Severity, and duration of influenza symptoms | 6 Months
  To characterize prevalence and duration of influenza symptoms before influenza and up to 6 months (acute phase and Long Flu).
Change in Health Related Quality of Life (HRQoL) using EQ-5D-5L | 6 Months
  To assess the change in HRQoL using EQ-5D-5L before COVID-19 or influenza and over a 6-month period following lab confirmed COVID-19 or influenza.
Change in Health Related Quality of Life (HRQoL) using WPAI:GH | 6 Months
  To assess the change in HRQoL using the Work Productivity and Activity Impairment Questionnaire: General Health (WPAI:GH) before COVID-19 or influenza and over a 6-month period following lab confirmed COVID-19 or influenza.
EQ-5D-5L Utility Index (UI) scores | 6 Months
  To estimate the EQ-5D-5L UI scores and their change over six months following lab confirmed COVID-19 or influenza.
Visual Analog Scale (VAS) scores | 6 Months
  To estimate the VAS scores and their change over six months following the lab confirmed COVID-19 or influenza.
Work Productivity and Activity Impairment (WPAI) scores | 6 Months
  To estimate the WPAI scores and their change over six months following the lab confirmed COVID-19 or influenza.

SECONDARY OUTCOMES:
Fatigue after COVID-19 or influenza | 6 Months
  To estimate the PROMIS questionnaire Fatigue short-form 8a score and its change over six months following lab confirmed COVID-19 or influenza.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591064